CLINICAL TRIAL: NCT04920890
Title: Effectiveness of Manual Therapy Combined With INDIBA Radiofrequency in the Recovery of Persistent Olfactory and Gustatory Alterations Post-COVID-19
Brief Title: Radiofrequency Intervention in Neurological Pathologies Post COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Gema Leon (Other)
Responsible Party: Principal Investigator, GEMA LEÓN BRAVO, Investigador principal, Clinica Gema Leon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ART-GLB-RF-COVID
Record Dates: First submitted 2021-05-26; First posted 2021-06-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Covid19; Neurological Injury; Olfactory Disorder; Gustatory Agnosia
Keywords: COVID-19; Multisystemic damage; Olfactory disorder; Gustatory agnosia; Radiofrequency Therapy
MeSH Terms: conditions — COVID-19; Trauma, Nervous System; Agnosia | interventions — Radiofrequency Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving radiofrequency treatment with manual therapy. (Experimental): Patients without previous pathology of any kind who have passed the Covid19 and have olfactory and gustatory sequelae; who will receive radiofrequency treatment with manual therapy.
  Interventions: Device: Radiofrequency therapy with manual therapy

INTERVENTIONS:
Device: Radiofrequency therapy with manual therapy — Monopolar Capacitive Resistive Radio Frequency at 448 kHz (INDIBA®) (RFMCR) with manual therapy.
  Other Names: INDIBA

SUMMARY:
The sequelae that occur in post-COVID-19 patients are multiple and, at a therapeutic level, these represent a new challenge within the general context of the pandemic that the world is suffering.

The virus has managed to end thousands of lives today and many other cases are being charged as directly responsible for a multiplicity of multi-system damages that need to be diagnosed and treated. Among the most relevant, are those that can affect to neurological levels in patients without previous pahologies, and in patients at risk who already had a pathology prior to infection.

On the other hand, signs and symptoms have been observed characteristic in the organ systems described above in post-contagion patients, directly associated with sequelae SARV-CoV2. The radio frequency (RF) of electromagnetic waves represents a technology of proven efficacy and safety in multiple fields of both human and veterinary medicine. These include neurological pathologies, and very especially those that affect the locomotor system. In therapeutics there are different RF modalities depending on the modality, polarity, type of signal and frequency, which in turn translate into different therapeutic profiles, clinical indications, efficacy and safety.

Among the RF technologies most used today and that have a greater scientific background, is the one known as Resistive Capacitive Monopolar Radio Frequency at 448 kHz (INDIBA®) (RFMCR). This study aims to assess the efficacy and safety of RFMCR in the treatment of neurological sequelae in patients presenting this type of pathologies that appear after contagion by COVID-19. Through this non-invasive technique, the investigators want to show that RF can help the physical rehabilitation of these patients through metabolic stimulation, increased vascularization and oxygenation of directly affected tissues, effects of deep hyperthermia generated by the interaction of the current with the treated biological substrate, as well as the activation of tissue regeneration, the result of subthermal action. It is thus intended to improve signs such as lung capacity, dyspnea, neuropathies and global muscle capacity, which are essential for the recovery of the post-COVID-19 patients.

The hypothesis of this study is that current post-COVID-19 treatments can be significantly improved in order to prevent complications and ensure the patients' well-being.

DETAILED DESCRIPTION:
The new post-pandemic era has left sequelae in patients who presented the signs and symptoms of SARS-CoV-2 and subsequently faced a positive for COVID-19. Such sequelae will be evident at various systemic levels of the affected patienta in the short, medium and long term future. One of these levels is neurological complications and injuries that have been documented throughout all scientific research since the beginning of massive infections worldwide.

SARS-CoV-2 is transmitted by penetrating the respiratory route (mostly), by fluid contact, and to a lesser extent, through the ocular pathway. In the field of neurology system, different forms of RF, nerve infiltrations, lymph node injuries, plantar fasciitis, spinal (peripheral) nerve disorders, etc. have been documented.

If the investigators focus on one of the most prevalent symptoms (those that affect the respiratory system), the bibliography that endorses that the RFMCR could improve has been referenced.

The aim of this study is to evaluate the efficacy of combined manual therapy and 448 kHz radiofrequency treatment in the recovery of persistent anosmia and ageusia in patients with post-COVID-19 sequelae. The work proposed here aims to demonstrate the advantages of establishing RF as an excellent treatment for post-COVID-19 sequelae, due to its ability to reinforce immune action, modulate the inflammatory response and activate cellular and tissue regeneration.

The specific objectives of this research work are:

1. To analyze the evolution of olfactory function using the Brief Smell Identification Test (BSIT) in patients treated with the combined protocol.
2. To evaluate the improvement in taste perception.
3. To determine the impact of treatment on quality of life.
4. To compare the results of taste and smell assessments between the different stages of treatment.
5. To examine the tolerance, safety and possible side effects of the combined treatment in post-COVID-19 patients.

REGULATIONS

1. This clinical study will be carried out in accordance with the protocol, the principles established in the current revised version of the Declaration of Helsinki (Fortaleza, 2013) and in accordance with the applicable regulatory requirements.
2. The researcher is aware, when signing the protocol, of the obligation to adhere to the instructions and procedures described in it, and will ensure that the established provisions are strictly adhered to.
3. The study will not begin until the approval of the Research Ethics Committee has been obtained.
4. The principal investigator is responsible for ensuring that this protocol, the informed consent document, and any other information that is presented or facilitated to the possible subjects is reviewed and approved by the CEI. The Researcher agrees to allow direct access to the REC to all relevant documents.

   INFORMED CONSENT.
5. In this case, patients must give their consent prior to being included in the study. The content and the procedure for obtaining it must be in accordance with all applicable legal requirements.
6. The investigator is responsible for obtaining the written informed consent of each patient participating in this study, after having explained in an understandable way, the nature, objectives, methods, expected benefits and possible risks of the study. The investigator must also explain to them that patients are completely free to refuse to participate in the study or to withdraw from it at any time, for whatever reason.
7. The study patients will give their consent, signing the corresponding model. For this purpose, each informed consent must be signed by both the investigator and the patient.

   CONFIDENTIALITY.
8. All information related to the study is considered confidential in compliance with the confidentiality and custody of the data collected, in accordance with the 3/2018 Law on the protection of personal data (LOPDGDD), (article 5). Article 5.1 .f) of the RGPD states that personal data will be treated in such a way as to guarantee confidentiality and integrity
9. In order to guarantee the confidentiality of the study data, only the main researcher and her team of collaborators will have access to it, the CEI and the pertinent health authorities.

FINANCING

1. The financing is assumed by the Gema León Physiotherapy and Rehabilitation Clinic. There is no direct economic consideration for this, although there is a dedication of time and work by the team of physiotherapists (social security, payroll, personal income tax, etc.) that is not economically remunerated and is assumed or absorbed this way. In addition, the RFMCR technology (equipment and accessories) will be provided by the company INDIBA S.A., through a temporary assignment without any financial compensation either from the Gema León Physiotherapy Clinic, or from any patient. The treatment of these is completely free for them.
2. The patient must travel to the clinic facilities and it is the researcher who will be responsible for the treatment in it.
3. No difficulties are foreseen in its performance since it will be carried out using a schedule adapted to the patient that allows the study to be monitored.

It is intended to carry out a longitudinal study with the participation of 10 patients with olfactory and gustatory alterations, who confirmed a positive test for COVID-19. The sample size for our study is large enough to detect a clinically important difference in the primary outcome (s). For this, the investigators reviewed references at the bibliographic level, in which paired studies obtained a statistically significant value, being able to support our study. If the sample size was insufficient but statistically significant, the investigators would resort to expanding the sample.

They will be evaluated at the beginning, a second evaluation after 3 weeks and a third final control after 12 sessions. A fourth evaluation will be carried out after the last and final evaluation, 6 weeks after finishing the treatment. Each of the participants will be informed of the study, the objective, its possible benefits and the side effects that could arise. A) Therefore, each patient must give their free and confirmed consent through signature. Among the items in the methodology, the following stand out:

Primary outcome: The assessment of smell was based on the short version of the Brief Smell Identification Test (BSIT). The short BSIT is a validated noninvasive 12-item test that uses odor strips of different characteristics to assess olfactory function.(15) A score of 0 (does not identify) or 1 (identifies odor but not as before) or 2 (identifies) is given for each item depending on whether the patient is able to identify the odor presented or not. Thus, any score below 16 out of 24 is considered to be altered smell.

Secondary outcome: Taste assessment was performed using the validated scale used in the article by Luigi Angelo Vaira et al. Four solutions of different tastes were provided: sweet, salty, sour and bitter. Taste scores ranged from 0 to 4, allowing patients to be classified into four categories: normal (score 4), mild hypogeusia (score 3), moderate hypogeusia (score 2), severe hypogeusia (score 1), and ageusia (score 0).

Tertiary outcome: To determine the social impact of loss of smell, the olfactory disorders questionnaire (sQOD-NS) was administered. The scores for the different questions range from 0 to 3, with 0 being none, 1 being a little, 2 being average and 3 being a lot. The total score for the questionnaire ranges from 0 (no impact on quality of life) to 21 (serious impact on quality of life).

The therapeutic protocol will be executed in the facilities of the Gema León Physiotherapy and Rehabilitation Clinic (Cordoba, Spain). Such RF therapeutic protocol will be implemented by application with an INDIBA® Activ device, whose function is to reduce inflammation, stimulate immunity and promote tissue regeneration. This will consist of a 45-minute treatment, composed by 15 minutes of treatment with the capacitive electrode and 30 minutes of the resistive electrode. A total of 12 sessions will be scheduled (two per week), and all processes will be documented from the beginning of therapy (the resources used will be provided by INDIBA and the Gema León Physiotherapy and Rehabilitation Clinic, whose supervision will be carried out by the direction of both).

Another variables which theyare gonna be take into accoont are sex, age, vaccination, number of days with symptoms and type of symptom.

The statistical analysis is based on variables of nominal type mostly, which are suitable for the Chi square test with a significance value of 95% for the results (p <0.05). However, if there are numerical data that must be compared between groups, the analysis will be used for ANOVA test with the same significance value for the comparison between results.

ELIGIBILITY:
Inclusion Criteria:

* Have passed the covid-19 disease without any previos pathology.
* Have olfactory and gustatory disorders one month later of COVID-19

Exclusion Criteria:

* Have passed the covid-19 disease with previous pathology, or not having passed the covid-19 disease.
* Have contraindications for the application of Indiba, such as pregnancy, pacemaker or thrombophlebitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Brief Smell Identification Test | 3 months
  A score of 0 is given (does not identify) or 1 (identifies odor but not the same as before) or 2 (identifies). Optimun value: 24
Validated Taste assesment from Luigi Angelo Vaira y cols. | 3 months
  Taste scores ranged from 0 to 4, allowing patients to be classified into four categories: normal (score 4), mild hypogeusia (score 3), moderate hypogeusia (score 2), severe hypogeusia (score 1), and ageusia (score 0). Optimal value: 16

SECONDARY OUTCOMES:
Questionnaire of olfactory disturbances (sQOD-NS) | 3 months
  It consists of 7 questions related to the quality of life and its relationship with food, anxiety, discomfort... The scores of the different questions vary from 0 to 3, with 0 being nothing, 1 being a little, 2 being average and 3 being a lot. The total score of the questionnaire ranges from 0 (no impact on quality of life) to 21 (serious impact on quality of life). Optimal value: 0

CONTACTS AND LOCATIONS:
Overall Officials: Gema León Bravo, Fisioterapia, Principal Investigator — Gema León Physiotherapy and Rehabilitation Clinic
Locations (1):
- Gema León Physiotherapy and Rehabilitation Clinic, Córdoba, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No
The request for the data will be studied and considered upon prior and justified request.